CLINICAL TRIAL: NCT06238102
Title: Psychiatric and Cognitive Assessment of Adult Patients With Hearing Impairment: the Impact on Quality of Life
Brief Title: Psychiatric and Cognitive Assessment of Adult Patients With Hearing Impairment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Yahia Hanafi mohamed, Resident doctor, Assiut University
Other Study IDs: Psychiatry and hearing
Record Dates: First submitted 2024-01-13; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: pure tone audiometry — measuring hearing impairment to select patients with hearing loss to evaluate who can this hearing impairment affects their quality of life

SUMMARY:
1. Assess the impact of hearing impairment on cognition
2. Evaluate the impact of hearing impairment on mental health
3. Evaluate the impact of hearing impairment on quality of life
4. Assess the relation between hearing loss and psychiatric disorder

DETAILED DESCRIPTION:
Hearing impairment is described as the partial or total loss of hearing ability. On the basis of the severity of the problem hearing impairment can be classified as mild, moderate, severe and profound. Age related hearing impairment is a very common disorder in older adulthood. It is considered as third most prevalent chronic health condition in people over 65 years of age. Hearing impairment in old age typically stems from some pathological changes inside the ear which are related to aging, it may lead to the impairment of low to high frequency hearing. This problem comes up with greater difficulty in listening process that significantly impairs person's ability to communicate with others, which in turn is a serious concern related to the mental health of individual.

It has been reported that adults with hearing loss tend to exhibit more symptoms of depression, anxiety, psychological distress, and emotional sensitivity as compared to people with normal hearing.

Hearing loss poses a serious risk to the mental well-being and overall quality of life in older adults. People may experience diminished self-esteem that in effect leads to the poor mental health and decline in psychological well-being.

Also, recent studies have demonstrated independent associations of hearing loss with incident dementia.

In Egypt such studies are lacking so investigators try to assess the impact of hearing loss on Psychiatry, Cognition and Quality of life by psychiatric interview, psychometric assessment , cognition assessment and quality of life assessment.

the aim is to evaluate the impact of hearing impairment on the above domains in Egypt

ELIGIBILITY:
Inclusion Criteria:

1. All patients diagnosed with hearing impairment
2. Age : 18 years and above
3. Gender: both sexes are included
4. willing to participate in the study
5. willing and able to provide informed consent

Exclusion Criteria:

1. Patients with intellectual disabilities
2. Patient with previous psychiatric and cognitive disorders
3. Patients with neurological diseases that affect hearing
4. Patients with history of chronic/ significant medical condition

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: people with hearing impairment (case) normal people without hearing impairment (control)
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the impact of hearing impairment on mental health by using Beck's depression scale | baseline
  we will use Beck's depression scale which is a 21-question multiple-choice self-report inventory, one of the most widely used psychometric tests for measuring the severity of depression. The highest possible total for the whole test would besixty-three.the lowest possible score for the test would be zero. High score indicate worse outcome
Evaluate the impact of hearing impairment on cognition by using montreal cognitive assessment | baseline
  we will use MoCA to assess cognition among people with hearing impairment. MoCA is widely used screening assessment for detecting cognitive impairment. It includes 11 questions with a maximum score of 30,a score of less than 24 indicates mild cognitive impairment
Evaluate the impact of hearing impairment on quality of life by using hearing handicap inventory for adults | baseline
  the Hearing Handicap Inventory for Adults (HHIA), is a 25-item self-assessment scale composed of two subscales (emotional and social/situational).this scale varies between 0 and 100; the social scale score can vary between 0 and 48 and the emotional scale can vary between 0 and 52. Higher values indicate a greater perception of the auditory handicap.

CONTACTS AND LOCATIONS:
Overall Officials: Hossam eldin khalifa, prof, Study Director — Assiut University

REFERENCES:
- [Background] Iwagami M, Kobayashi Y, Tsukazaki E, Watanabe T, Sugiyama T, Wada T, Hara A, Tamiya N. Associations between self-reported hearing loss and outdoor activity limitations, psychological distress and self-reported memory loss among older people: Analysis of the 2016 Comprehensive Survey of Living Conditions in Japan. Geriatr Gerontol Int. 2019 Aug;19(8):747-754. doi: 10.1111/ggi.13708. Epub 2019 Jun 24. PMID 31237108
- [Background] Shear MK, Vander Bilt J, Rucci P, Endicott J, Lydiard B, Otto MW, Pollack MH, Chandler L, Williams J, Ali A, Frank DM. Reliability and validity of a structured interview guide for the Hamilton Anxiety Rating Scale (SIGH-A). Depress Anxiety. 2001;13(4):166-78. PMID 11413563
- [Background] Lin FR, Metter EJ, O'Brien RJ, Resnick SM, Zonderman AB, Ferrucci L. Hearing loss and incident dementia. Arch Neurol. 2011 Feb;68(2):214-20. doi: 10.1001/archneurol.2010.362. PMID 21320988
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Isaacson B. Hearing loss. Med Clin North Am. 2010 Sep;94(5):973-88. doi: 10.1016/j.mcna.2010.05.003. PMID 20736107
- [Background] Newman CW, Weinstein BE, Jacobson GP, Hug GA. Test-retest reliability of the hearing handicap inventory for adults. Ear Hear. 1991 Oct;12(5):355-7. doi: 10.1097/00003446-199110000-00009. PMID 1783240